CLINICAL TRIAL: NCT04267666
Title: Comparative Study of Inspiratory Muscle Strength Training and Incentive Spirometer on Ventilatory Function in Postmenopausal Asthmatic Women
Brief Title: Inspiratory Muscle Strength Training and Incentive Spirometer on Postmenopausal Asthmatic Women
Acronym: training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoU9
Record Dates: First submitted 2020-01-31; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Asthmatic; Postmenopausal Symptoms
Keywords: Inspiratory; Spirometer; Postmenopausal; asthma
MeSH Terms: conditions — Asthma; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: inspiratory muscle training in the form of: Inspiratory threshold muscle trainer in addition to traditional chest physical therapy intervention (Deep breath, cough training)
Who Masked: Outcomes Assessor
Masking Description: Participants were assigned randomly used sealed envelope into two groups (A&B) equally in number.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Strength Training (Experimental): in the form of: Inspiratory threshold muscle trainer in addition to traditional chest physical therapy intervention (Deep breath, cough training)
  Interventions: Other: Inspiratory muscle trainer device
- Incentive Spirometer (Experimental): incentive spirometer, three sessions per week for six weeks
  Interventions: Device: incentive spirometer

INTERVENTIONS:
Device: incentive spirometer — Patient had to produce a high inspiratory pressure. The ball serves as visible feedback of the inspiratory flow and indicates the obtained flow on a calibrated scale on the transparent cylinder of the spirometer. If the patient flows greater than 300 milliliters per second, the float ball in first chamber will rise. As patient flow increases to 600 milliliters per second the second ball float will rise. If the patient flow exceeds 900 milliliters per second all three will be suspended. Patient should encourage holding the balls up for a few seconds
  Arms: Incentive Spirometer
Other: Inspiratory muscle trainer device — The threshold trainer is a small plastic handheld device supplied by respironics. It includes a mouthpiece and a calibrated spring loaded valve. The valve controls a constant inspiratory pressure training load and the patient must generate the inspiratory pressure in order for the inspiratory valve to be opened and allow inhalation of air.
  Arms: Inspiratory Muscle Strength Training

SUMMARY:
Objective: To compare the effectiveness of inspiratory muscle training (IMT) and incentive spirometer on ventilatory functions in post-menopausal asthmatic women. Participants and methods: A total of forty postmenopausal women suffering from asthma, their ages ranged from 50 to 60 years old, and their body mass index of the patient don't exceed 30kg/m2. They were recruited from patient chest clinic in Kasr -El- Ainy Teaching Hospital, Cairo University, Egypt.

DETAILED DESCRIPTION:
They signed a consent form, confidentiality was assured. They assigned into two groups (A) who received inspiratory muscle training in the form of: Inspiratory threshold muscle trainer in addition to traditional chest physical therapy intervention (Deep breath, cough training) while patients in group (B): received traditional chest physical therapy intervention and incentive spirometer, three sessions per week for six weeks. Patients in both groups were assessed before treatment (pre-training) then after treatment (post-training) (after 6 weeks) to measure lung functions using electronic spirometer. The training program was carried in the duration from January 2019 to July 2019.

ELIGIBILITY:
Inclusion Criteria:

* Forty postmenopausal women suffering from asthma
* Their ages were ranged from 50 to 60 years,
* their body mass index (BMI) don't exceed 30kg/m2.
* All participants were asthmatic patient
* clinically and medically stable cases

Exclusion Criteria:

* participant who had chest infection,
* malignant diseases,
* Patients with chest trauma.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Electronic Spirometer (VIASYS- Health Care Microlab) | 6 weeks
  It was used for ventilatory functions measurement Ventilatory,reported as a number in liters (L).
FVC (Forced vital capacity) | 6 weeks
  is one of the most useful tests to assess the overall ability to move air in and out of the lungs (ventilation). This is the maximum amount of air that can be forcefully and rapidly exhaled after a deep breath (maximal inspiration),reported as a number in liters (L)
FEV1 (Forced expiratory volume) | 6 weeks
  is the volume of air forcibly exhaled in one second during the FVC test,reported as a number in liters (L)
MVV (Maximum voluntary ventilation) | 6 weeks
  is the maximum air, which can be expired in a minute by deepest and fastest breathing, reported as a number in liters (L)

SECONDARY OUTCOMES:
Body mass index | 6 weeks
  It was used for measuring the weight and height of each patient to calculate the body mass index. BIM=weight (Kg) / height (m2).

CONTACTS AND LOCATIONS:
Overall Officials: ghada eb elrefaye, professor, Principal Investigator — Department of Physical Therapy for Women's Health, Cairo University, Egypt.
Locations (1):
- Ghada Ebrahim Elrefaye, Giza, Dokki, Egypt